CLINICAL TRIAL: NCT02353897
Title: An Assessment of Patient and Physician's Satisfaction After a Long Term Treatment of Glabellar Lines With Dysport®.
Brief Title: Patient and Physician's Satisfaction After a Long Term Treatment of Glabellar Lines With Dysport®
Acronym: APPEAL
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: Y-79-52120-201
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Glabellar Lines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to look at patient and physician satisfaction of long term Glabellar lines (GL) treatment with Dysport in a real life setting. It will also allow better understanding of what patients expect from the treatment, and the injection practices used by doctors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with moderate to severe GL naïve of any type of aesthetic treatment/procedure (invasive and non-invasive) for GL who provided written informed consent to take part.
* Patient who has prior to and independent of the study decided to undergo long term treatment of GL only (at least three cycles).
* Patient able to comply with the protocol (completion of web questionnaires).
* Patient whom physician intended to treat with Dysport independent of participation in the study.

Exclusion Criteria:

* Patient already included in this study.
* Participation in an interventional trial within 30 days prior to study entry.
* Patient who is at risk in terms of precautions, warnings, and contraindication (follow local Summary of Product Characteristics (SmPC) of Dysport).
* Female patient who is pregnant, nursing or planning a pregnancy during the study.
* Hypersensitivity to Dysport® or to its excipients.
* Presence of infection at the proposed injection sites.
* Presence of myasthenia gravis, Eaton Lambert syndrome or amyotrophic lateral sclerosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Private practices and clinics
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
To assess patient satisfaction regarding GL after three injection cycles of Dysport. | Within 3 weeks ±7 days of visit 3
  Assessed by patient auto questionnaire completion

SECONDARY OUTCOMES:
To describe patient individual expectations. | Within 3 weeks ±7 days of visit 1 and 2
  Assessed by patient auto questionnaire completion
To assess patient satisfaction after one and two injection cycles of Dysport. | Within 3 weeks ±7 days of visit 1 and 2
  Assessed by patient auto questionnaire completion
To describe factors associated with patient satisfaction such as attractiveness, self-esteem, self-perceived age, desire to receive another injection. | Within 3 weeks ±7 days of visit 1 and 2
  Assessed by patient auto questionnaire completion
To assess the GL severity (at rest and maximum frown) as per usual practice. | Baseline (visit 1) and visit 3
  Physician assessment using GL severity scale
To assess physician satisfaction after one and three injection cycles of Dysport. | Visit 1 follow up visit and visit 3 follow up visit (if performed)
  5 point Likert scale
To describe Dysport injection practices: muscles injected, total injected units, total volume injected, number of injection points and interval between injections. | From visit 1 until the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (14):
- Australia (2):
  - ERASE, Malvern
  - SouthDerm, Sydney
- Clinica Laura Bariquelo Buratini, Botucatu, Brazil
- Czechia (2):
  - Estetická Dermatologie, Brno
  - BcD Clinic s.r.o., Prague
- Laser Center DARUS, Almaty, Kazakhstan
- Dr Haddad Clinics, Beirut, Lebanon
- Russia (5):
  - Centre of Aesthetic Medicine "Chistie prudi", Moscow
  - Preventive Medicine Clinic "Vallex M", Moscow
  - Plastic Surgery Institute, Moscow
  - FI IF & TC & apos; Eye microsurgery & apos, Novosibirsk
  - Clinic of Aesthetic Medicine, Saint Petersburg
- Kocaeli University School of Medecine Umuttepe, Kocaeli, Turkey (Türkiye)
- Clinic of Aesthetic medicine "Ankor", Kyiv, Ukraine

REFERENCES:
- [Derived] Gubanova E, Haddad Tabet M, Bergerova Y, Moiseieva O, Chemeris A, Sanches E, Sharova A, Rodriguez Pose L, Raymond R, Prygova I, Carlisle I. Assessment of Subject and Physician Satisfaction after Long-Term Treatment of Glabellar Lines with AbobotulinumtoxinA (Dysport(R)/Azzalure(R)): Primary Results of the APPEAL Noninterventional Study. Aesthetic Plast Surg. 2018 Dec;42(6):1672-1680. doi: 10.1007/s00266-018-1200-4. Epub 2018 Aug 17. PMID 30120518